CLINICAL TRIAL: NCT00019578
Title: Phase I Pilot Study of Stereotaxic Radiosurgery in Patients With Intracranial Neoplasms
Brief Title: Stereotactic Radiosurgery in Treating Patients With Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990011; 99-C-0011; CDR0000066758; NCT00001791 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2012-03

CONDITIONS: Adult Central Nervous System Germ Cell Tumor; Adult Malignant Meningioma; Adult Medulloblastoma; Adult Noninfiltrating Astrocytoma; Adult Oligodendroglioma; Adult Craniopharyngioma; Adult Meningioma; Brain Metastases; Adult Ependymoma; Adult Pineal Parenchymal Tumor; Adult Brain Stem Glioma; Adult Infiltrating Astrocytoma; Mixed Gliomas; Stage IV Peripheral Primitive Neuroectodermal Tumor
Keywords: adult brain stem glioma; adult brain tumor; adult central nervous system germ cell tumor; adult craniopharyngioma; adult ependymoma; adult infiltrating astrocytoma; adult malignant meningioma; adult medulloblastoma; adult meningioma; adult noninfiltrating astrocytoma; adult oligodendroglioma; adult pineal parenchymal tumor; adult solid tumor; body system/site cancer; brain metastases; brain tumor; cancer; central nervous system cancer; genetic condition; metastatic cancer; mixed gliomas; site, metastatic cancer; solid tumor; stage IV peripheral primitive neuroectodermal tumor; stage/type, adult brain tumor; unclassified/other cancer
MeSH Terms: conditions — Meningioma; Medulloblastoma; Oligodendroglioma; Craniopharyngioma; Brain Neoplasms; Ependymoma; Pinealoma; Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Neoplasms; Central Nervous System Neoplasms; Genetic Diseases, Inborn; Neoplasm Metastasis

INTERVENTIONS:
Procedure: Sterotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. PURPOSE: Phase I trial to study the effectiveness of stereotactic radiosurgery in treating patients who have brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Establish stereotaxic radiosurgery as a treatment technique at the National Institute of Health in patients with intracranial neoplasms.

II. Assess the response rate, local control, time to progression, pattern of failure, and magnetic resonance spectrographic data following this therapy in these patients.

PROTOCOL OUTLINE: All patients undergo stereotaxic head frame placement, followed by stereotaxic radiosurgery on day 1. The dosage of radiation therapy administered is dependent on the tumor diameter.

Patients are followed at 2 and 6 weeks and then every 3 months for 5 years.

PROJECTED ACCRUAL:

Up to 30 patients will be accrued for this study within 7-10 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven intracranial tumor OR Pathologically confirmed cancer with metastases to the brain OR Newly discovered brain lesions that are amenable to stereotaxic biopsy No more than 3 measurable tumors Only 1 tumor more than 3 cm in diameter that requires radiosurgery allowed No tumor more than 4 cm in diameter No tumor that involves more than 50% of the brain stem --Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Concurrent corticosteroids allowed Radiotherapy: Prior cranial radiotherapy allowed Surgery: Radiosurgery to other nonstudy intracranial lesions allowed Prior biopsy and/or subtotal or near-total resection allowed --Patient Characteristics-- Age: 18 and over Performance status: Karnofsky 70-100% OR ECOG 0-2 Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count at least 500/mm3 Hemoglobin at least 10 g/dL Platelet count at least 50,000/mm3 Hepatic: SGOT or SGPT no greater than 2.5 times upper limit of normal (ULN) PT and PTT no greater than 1.5 times ULN No clinically significant hepatic dysfunction Renal: Creatinine no greater than 1.3 times ULN Cardiovascular: No clinically significant cardiac dysfunction Pulmonary: No clinically significant pulmonary dysfunction Other: Not pregnant or nursing Negative pregnancy test No clinically significant systemic illness or serious infection that would preclude study compliance No other organ dysfunction that would preclude study compliance No history of psychiatric disease No allergy to contrast agent Papilledema and motor or sensory deficits allowed No contraindications to MRI (e.g., aneurysm clip, implanted neural stimulator, implanted cardiac defibrillator, cochlear implant, ocular foreign body or implant, or insulin pump)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian G. Fuller, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Radiation Oncology Branch, Bethesda, Maryland, United States